CLINICAL TRIAL: NCT05811767
Title: Ergonomic Exposure in Relation to Physical Capacity and Its Effect on Work Ability and Musculoskeletal Pain in the Oldest Group of Workers - The Esbjerg Cohort
Brief Title: The Esbjerg Cohort - A Cross-sectional Study About Work Ability and Musculoskeletal Pain in 55 to 70 Years Old Workers
Status: Completed | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: esbjerg_cohort
Record Dates: First submitted 2023-03-16; First posted 2023-04-13 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Work Ability; Occupational Health; Physical Capacity; Occupational Exposure
Keywords: Work ability; Senior workers; Physical capacity; Musculoskeletal pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Nutrition Surveys

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A blood test examinate for cholesterol (total cholesterol, HDL and LDL) and D-vitamin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Esbjerg Cohort: This is a cross-sectional study and therefore there is no intervention to describe. The study consist only of tests, questionnaires and a blood test. See the elements under outcomes measures.
  Interventions: Other: Health Examination

INTERVENTIONS:
Other: Health Examination — The study is a cross-sectional study and therefore there is no intervention. The study consist only of tests, questionnaires and a blood test. See the elements under outcomes measures.

SUMMARY:
The overall aim of this study is to investigate how work with physical demands affects the physical capacity, work ability, labor market affiliation, pain and self-reported health in the oldest group of workers.

Following research questions are to be answered:

1. How high physical work demands affects muscle strength in 55-70-year-old workers and how obesity in combination with high physical work exposure influences muscle strength, work ability, cardiac function, and self-reported health?
2. Which parameters are important for work ability and how does the exposure of high physical workload affect the work ability over time in 55-70-year-old workers?
3. By exploring the underlying mechanism of pain among 55+ year old workers, how is pain associated with work ability, BMI and physical capacity?

DETAILED DESCRIPTION:
This study is a population-based cross-sectional study conducted in the municipality Esbjerg, Denmark. This study wants to investigate how ergonomic exposure in relation to physical capacity has an effect on work ability and musculoskeletal pain in workers between 55 and 70 years old. This Ph.D. is a clinical study including physical tests, questionnaires, and long-term evaluation of work ability. The study population consists of 336 citizens divided into 12 groups stratified for gender, age (< 60 years, 60-64 years and above 64 years) and occupational group (white-collar or blue-collar worker).

The study population will be recruited to uncover the physical workload among citizens 55+ years and compare the physical work demands to their health status, pain and physical capacity. The intention is to provide knowledge of the consequences of high physical workload on the musculoskeletal system in the oldest group of workers. This knowledge is necessary for better treatment and counseling to the oldest group of workers and for improved guidelines on how to optimize the balance between the physical work demands and the capacity of the workers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women born between 1952 and 1966
* Living in the Esbjerg municipality
* Able to write, read and understand Danish

Exclusion Criteria:

* Injuries to arms or legs (e.g arm in plaster, acute trauma on ACL)
* Just had a surgery (e.g an operation in the abdominal region or in the brain)

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Citizens between 55 and 70 years old living in the Esbjerg municipality.
Sampling Method: Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Work Ability | Baseline
  Measured with Work Ability Index (WAI), which is a questionnaire, measuring seven items to assess the workers work ability

SECONDARY OUTCOMES:
Height | Baseline
  Measured in centimeters
Weight | Baseline
  Measured in kilograms
Body Mass Index (BMI) | Baseline
  Calculated by kg/m^2
Waist-to-hip ratio | Baseline
  Measured in centimeters between the hip and the waist
Blood pressure | Baseline
  Both diastolic and systolic
Pressure Pain Threshold | Baseline
  A part of the quantitative sensory testing battery. Measured with an algometer three times on thenar eminence at the non-dominant hand and at tibialis anterior on the non-dominant leg
Warm and cold detection threshold | Baseline
  A part of the quantitative sensory testing battery. Measured with a TSA 2001-II machine on thenar eminence at the non-dominant hand. The temperature rises and falls three times each with 1°C/s. The participant press a button, when they feel a change in temperature.
Heat and cold pain threshold | Baseline
  A part of the quantitative sensory testing battery. Measured with a TSA 2001-II machine on thenar eminence at the non-dominant hand. The temperature rises falls three times each with 1°C/s. The participant press a button, when they detects pain.
Temporal summation | Baseline
  A part of the quantitative sensory testing battery. Measured with a TSA 2001-II machine. Ten brief repetitive heat pulses at thenar eminence on both hands. There the participant rates the second pain approximately one second after each stimulus.
Conditioned pain modulation | Baseline
  A part of the quantitative sensory testing battery. Two separate stimuli were used. A test stimulus and a conditioning stimulus. The test stimulus consisted of pressure pain threshold measurements as described above. The test stimulus was performed on the non-dominant hand at the thenar eminence and tibialis anterior before and immediately after the conditioning stimulus, with one minute between the two test sides. The conditioning stimulus was a cold pressor test which consisted of cold water (10°C) immersion of the hand on the dominant side down to the wrist for a duration of two minutes.
Physical Activity | Baseline
  Measured with The international Physical Activity Questionnaire (IPAQ), which is a 27-item self-reported questionnaire about physical activity for the last seven days at work and in spare time.
Musculoskeletal pain | Baseline
  Measured with Nordic Musculoskeletal Questionnaire (NMQ). NMQ consist of a generally questionnaire to asses musculoskeletal disorders in nine anatomical region (ex. Shoulder, low back and knee). In addition, NMQ contains special questionnaires for low back, neck and shoulder symptoms to probe these areas more deeply. In this questionnaire, there have been an extension in the special questionnaires to all nine anatomical regions.
Additionally questions about ergonomic and pain | Baseline
  In addition to the standardized questionnaires described above, an extra questionnaire with further questions about the participant's ergonomics in their work and more generally about their pain on a scale from zero to ten.
30-seconds sit to stand test | Baseline
  Used to test the strength and endurance in the legs. Its measures how many times the participant can get up from a chair in 30 seconds.
Balance test | Baseline
  Performed with a one-leg balance test. It measure how low the participant can stand on one leg with the arms on the waist.
Stair climb test | Baseline
  Measures functional strength, balance and agility. The participant must climb up and down a flight of stairs as quickly as possible.
Maximal aerobic capacity (VO2 max) | Baseline
  Measured with a sub maximal treadmill exercise test, known as Astrand 6 minute cycle test
Isokinetic muscle strength in the shoulder | Baseline
  Measured with a Biodex System 4 dynamometer. The dominant shoulder is tested. The participant makes an abduction and adduction as fast and powerful they can. The test is performed three times with 15 seconds rest between the tests.
Isometric muscle strength in the shoulder | Baseline
  Measured with a Biodex System 4 dynamometer. An isometric contraction in abduction in the dominant shoulder. The participant keeps the tension in 3-5 seconds with 40 seconds break between each test.
Isokinetic muscle strength in the knee | Baseline
  Measured with a Biodex System 4 dynamometer. The non-dominant knee is tested. The participant makes an extension and flexion as fast and powerful they can. The test is performed three times with 15 seconds rest between the tests.
Isometric muscle strength in the knee | Baseline
  Measured with a Biodex System 4 dynamometer. An isometric contraction in extension in the non-dominant knee. The participant keeps the tension in 3-5 seconds with 40 seconds break between each test.
Handgrip strength | Baseline
  Performed with a JAMAR hand dynamometer. The participant press the dominant hand as hard as they can for three to five seconds. The test is performed three times with 15 seconds break between each test.
Psychosocial work environment | Once after baseline
  Measured with the Danish Psychosocial Work Environment Questionnaire (DPQ). DPQ is a questionnaire used to evaluate the physical work environment (11). It contains 38 themes regarding to physical work environment within five overall dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ejstrup, MSc, Principal Investigator — The Hospital South West Jutland, University hospital of Southern Denmark
Locations (1):
- The Hospital South West Jutland, University hospital of Southern Denmark, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is under current Danish law not feasible.